CLINICAL TRIAL: NCT00004002
Title: Phase I Trial of PS-341 in Advanced Cancers
Brief Title: PS-341 in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067212; NYU-9909; NCI-T99-0047
Record Dates: First submitted 1999-11-01; First posted 2004-04-12 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2005-09

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bortezomib

INTERVENTIONS:
Drug: bortezomib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of PS-341 in treating patients who have advanced solid tumors or lymphoma that have not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the dose-limiting toxicity and maximum tolerated dose of PS-341 in patients with advanced solid tumors or lymphoma. II. Evaluate the pharmacodynamics of this drug by measuring 20S proteasome inhibition in these patients. III. Assess changes in P53 or P27, and possibly E2F-1 and cyclin E, in patients with lymphoma in response to this drug. IV. Evaluate objective tumor response to this drug in these patients. V. Evaluate the relationship between toxicity and 20S proteasome inhibition in blood and in accessible tumor tissue in these patients. VI. Evaluate response to treatment with this drug in patients with measurable or evaluable disease.

OUTLINE: This is a dose-escalation, multicenter study. Patients receive PS-341 IV on days 1 and 4. Treatment repeats every 14 days for at least 2 courses in the absence of unacceptable toxicity or disease progression. Patients with stable or responding disease may receive additional courses at the discretion of the treating physician. Cohorts of 3-6 patients receive escalating doses of PS-341 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 6 patients experience dose-limiting toxicity. Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A maximum of 27 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid tumor or lymphoma that has failed standard therapy and no standard options available No leukemia or myeloma CNS lesions allowed if adequately treated by surgery and/or radiotherapy and symptomatically stable on maintenance glucocorticoids and not requiring anticonvulsants for at least 3 months

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT no greater than 2.5 times upper limit of normal Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No acute ischemia or significant conduction abnormality (i.e., bifascicular block or 2nd or 3rd degree AV blocks) Other: No other serious medical or psychiatric illness Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow transplantation with high-dose chemotherapy or radiolabeled monoclonal antibody therapy for lymphoma patients Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas) Endocrine therapy: See Disease Characteristics Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: At least 2 weeks since prior major surgery Other: See Disease Characteristics No concurrent antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health
Locations (5):
- United States (5):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York

REFERENCES:
- [Result] Hamilton AL, Eder JP, Pavlick AC, Clark JW, Liebes L, Garcia-Carbonero R, Chachoua A, Ryan DP, Soma V, Farrell K, Kinchla N, Boyden J, Yee H, Zeleniuch-Jacquotte A, Wright J, Elliott P, Adams J, Muggia FM. Proteasome inhibition with bortezomib (PS-341): a phase I study with pharmacodynamic end points using a day 1 and day 4 schedule in a 14-day cycle. J Clin Oncol. 2005 Sep 1;23(25):6107-16. doi: 10.1200/JCO.2005.01.136. PMID 16135477